CLINICAL TRIAL: NCT03505866
Title: Investigating the Impact of Community Home-based Care Intervention on Mental Health Outcomes and Anti-retroviral Therapy Adherence in People Living With HIV
Brief Title: Community Home-based Care Intervention and Its Health Outcome in HIV-positive People
Acronym: HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrated Development Foundation Nepal (Other)
Collaborators: Tokyo University (Other)
Responsible Party: Principal Investigator, Khem Narayan Pokhrel, Research and Program Development Advisor, Integrated Development Foundation Nepal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1523
Record Dates: First submitted 2018-04-01; First posted 2018-04-23 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Human Immunodeficiency Virus; Depression; Stress; Anxiety; Quality of Life
Keywords: HIV; Anti-retroviral therapy; Intervention; Mental Health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The intervention was started in February and March, 2015 and was completed six month later. The program comprises of psychosocial support/peer counseling, ART adherence support and counseling, basic health care, and referral for further care. The support team comprises of a community health worker, a trained HIV-positive person, and a social worker.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mutual support groups of HIV (Other): HIV-positive people who did not enroll in a community home-based care intervention and receiving regular HIV services and support from mutual support groups of HIV
  Interventions: Behavioral: Community home-based care intervention

INTERVENTIONS:
Behavioral: Community home-based care intervention — HIV-positive people who received community home-based care intervention on a monthly basis for six months after they enrolled in the program.

SUMMARY:
An intervention study was designed to examine the impact of impact of community home-based care intervention on mental health and treatment outcome in HIV-positive people. The intervention comprised a home-based counseling on anti-retroviral therapy (ART) adherence, psycho social support, basic health care services at the home of HIV-positive people. The intervention started in March, 2018 and completed in August 2018. The major measurements of the interventions were ART adherence, status of depression, anxiety, and stress levels.

DETAILED DESCRIPTION:
HIV continues to be a global health problem, particularly mental health status and non-adherence to ART remains challenges in people living with HIV (PLHIV) in low- and middle-income countries. Mental health disorders, particularly those who experience depression and anxiety may endure poor satisfaction or trust to the treatment, leading to non-adherence to ART. Also, those, who have high level of perceived stress may not seek adequate social support from care givers and service providers, that may worsen their ART adherence. Substance use also induces poor coping skills and poor dependence on treatment.

HIV positive people also experience co-occurring mental health disorders and substance use. For instance, those who experienced depression are more likely to develop the risk of substance use compared to those who did not experience depression. Similarly, those who engage in substance use such as amphetamine, cocaine, and opioid may develop the risk of chronic stress. However, evidence is limited about the prevalence of co-occurring pattern of these conditions on ART adherence among them worldwide.

Psychosocial support may be an integral part of HIV care and support to meet the mental health needs of people living with HIV. To address the need for psychosocial support, WHO provided the guideline to manage their psychological and social problems. The guideline recommends that HIV-positive people, their families, and caregivers receive psychosocial support at family, community, and health facility level. It also suggests that psychosocial support should be an integral part of care and support framework for HIV services.

Community and home-based care program is designed as a WHO framework for providing psychosocial support and basic health care to PLHIV. According to this framework, it is defined as any form of care given to ill people in their homes. Such care includes physical, psychosocial, palliative, and spiritual activities. The goal of this program is to provide hope through high-quality and appropriate care that helps ill people and families to maintain their independence and achieve the best possible QOL. The program may incur low cost or can be sustainable strategy for providing comprehensive services at the home of PLHIV.

In Nepal, 23 non-governmental organizations (NGOs) provide care and support services through community home-based care program in Nepal. The program comprises psychosocial support, ART adherence and support, peer counseling, basic health care, referral for further care. However, little is known about the role of community home-based care program in reducing depression, anxiety and high stress level among people living with HIV in the country. In addition, they receive peer counseling about their substance use, however, no study examined the role of such intervention to reduce substance use. Also, the program comprises ART support and counseling to HIV positive people and their family, no study has examined its effect on non-adherence to ART. This study is aimed to assess the impact of community home based care program on depressive symptoms, anxiety, high stress, and substance use and non-adherence to ART.

A intervention study was conducted among 682 PLHIV in Nepal. Among them, 344 participants were assigned for community and home-based care intervention and 338 were assigned for control. Baseline information was collected including sociodemographic characteristics, HIV/AIDS clinical staging, depressive symptoms, anxiety, and stress scores, substance use. Depressive symptoms were measured using center for epidemiological study depression scale (CESD). Anxiety was measured with composite international diagnostic interview-short form (CIDI-SF). Perceived Stress Scale measured stress scores. ART non-adherence was measured if participants missed at least two pills in past months.

After six months, a follow up survey was done and collected the information as baseline. The analysis was done with mainly three strategies. First, the associations of independent and combined mental health disorders and substance use with non-adherence to ART were examined using logistic regressions stratified by gender. Separate models for generalized estimating equation (GEE) were applied to measure the effect of community home-based care intervention on various outcomes. Two models for GEE were developed. First, the effect of community home-based care intervention on depression, anxiety, high stress and substance use were assessed. Second GEE model examined the effect of intervention on non-adherence to ART. In all GEE multivariable models, age, gender, marital status, education, employment, HIV/AIDS clinical staging, and presence of physical symptoms were controlled.

Keywords: Mental health, Anti-retroviral therapy adherence, intervention, Nepal

ELIGIBILITY:
Inclusion Criteria:

1. HIV-positive people who did not enroll in a community home-based care program before the baseline data collection for intervention. Those who were referred by an ART center or a voluntary counseling and testing center for care and support services
2. Those who were diagnosed as HIV-positive within five years of baseline data collection and living in the selected districts for at least one year
3. Those who received pre-ART counseling services and were receiving ART for at least one year
4. Those who voluntarily agreed to enroll in a community home-based care program and received intervention after the baseline study.

Exclusion Criteria:

The exclusion criteria were being hospitalized for an intensive care at the time of data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Depression | 6 months
  Depression was measured using a Center for Epidemiologic Studies Depression (CESD) scale. This scale consists of 20 items that are designed to measure the participant's experience of depressive symptoms in the past week of data collection. The total scores range from 0 to 60, and, a cut off point was set as scores ≥ 16 designating the occurrence of depressives symptoms.
Anti-retroviral therapy non-adherence | 6 months
  Adherence to anti-retroviral therapy was measured using AIDS Clinical Trial Group Questionnaires. The questionnaires are designed to measure non-adherence whether the HIV-positive person missed at least one dose of anti-retroviral therapy in the past month of the data collection. The questionnaire assess
Anxiety | 6 months
  Anxiety was measured anxiety using Composite International Diagnostic Interview Short-Form (CIDI-SF) the scale use nine screening stem questions that were designed to measure the episodes of anxiety and their control over their worries and anxious state.
stress | 6 months
  Stress was in the past month using the Perceived Stress Scale (PSS). It consists of 10 items with scores ranging from "0" (never) to 4 (very often). The total score ranges from 0-40. Higher stress scores indicate high level of stress.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pokhrel KN, Sharma VD, Pokhrel KG, Neupane SR, Mlunde LB, Poudel KC, Jimba M. Investigating the impact of a community home-based care on mental health and anti-retroviral therapy adherence in people living with HIV in Nepal: a community intervention study. BMC Infect Dis. 2018 Jun 7;18(1):263. doi: 10.1186/s12879-018-3170-1. PMID 29879916